CLINICAL TRIAL: NCT01360606
Title: A Phase I Study of Stereotactic Body Radiation Therapy (SBRT) for Liver Metastases
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Liver Mets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susannah Ellsworth (Other)
Responsible Party: Sponsor-Investigator, Susannah Ellsworth, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 09-051
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Liver Metastases
Keywords: Stereotactic Body Radiation Therapy (SBRT); standard uptake value (SUV)
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SBRT (Other)
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT:
  Patients will receive one of the following radiation regimens:
  * 50 Gy in 5 fractions (10 Gy/fx) delivered over a 2-week period.
  * 60 Gy in 5 fractions (12 Gy/fx) delivered over a 2-week period.
  * 75 Gy in 5 fractions (15 Gy/fx) delivered over a 2-week period.
  Other Names: CyberKnife; Trilogy; True Beam; Radiosurgery

SUMMARY:
This is a phase I dose escalation study. Dose escalation will be via the traditional "up and down" scheme. SBRT:

Patients will receive one of the following radiation regimens:

* 50 Gy in 5 fractions (10 Gy/fx) delivered over a 2-week period.
* 60 Gy in 5 fractions (12 Gy/fx) delivered over a 2-week period.
* 75 Gy in 5 fractions (15 Gy/fx) delivered over a 2-week period.

DETAILED DESCRIPTION:
Prior to enrollment all patients will be evaluated with a physical exam, review of pathology and laboratory values to confirm diagnosis, and baseline imaging studies.

Accelerator

Physicians will treat with a stereotactic radiosurgery system using 6MV photons to deliver stereotactic body radiotherapy.

Doses

Patients will receive a total dose ranging from 50-75 Gy in 5 fractions (10-15 Gy/fx). Dose escalation will be via the traditional "up and down" scheme.

In determining the radiation dose and fractionation scheme for this protocol, we used the linear-quadratic formalism for radiation cell killing to "equate" schemes that vary the dose/fraction and number of fractions. This concept of biologically equivalent dose (BED) states that the total effect is given by:

nd x (1 + d/(alpha-beta ratio))

where n is the # of fractions and d is the dose/fraction. The "alpha-beta ratio" characterizes the radiation response of a particular tissue; a higher value is indicative of a tissue that responds acutely to the effects of radiation. Due to their highly proliferative nature, most tumors fall into this category.

This final dose scheme (total dose 75 Gy) is biologically equivalent to the previously studied doses in the literature (60 Gy in 3 fractions), meaning the first two sets of patients will be treated to a radiobiologically smaller (and likely safer) dose. We would favor treating in five fractions, as opposed to three, to allow more repair of normal tissue, reoxygenation of tumor cells, and redistribution of tumor cells to more radiosensitive parts of the cell cycle. Using a smaller fraction size, 10-15 Gy compared to 20 Gy, will also help reduce late effects of radiation therapy. SBRT treatment will be given on an every other day schedule, excluding weekends. The prescription dose will be prescribed to the isodose line best encompassing the planning target volume (PTV) depending on the volume of tumor (HCC).

Localization, immobilization, and simulation

Within 5 - 10 days after fiducial placement, pPatients will undergo 4D FDG-PET/CT simulation with the goal of evaluating tumor motion to allow for gated treatment when indicated. This goal will be accomplished by using the Real-time Position Management (RPM) system (Varian Medical Systems, Palo Alto, CA) to create a retrospective 4D CT scan. Following the institutional protocol, a helical CT scan and a 4D positron emission tomography (PET) scan with a patient with body immobilization device will be acquired. A patient will not eat or drink anything for four hours before the PET scan. Before the PET scan, blood sample will be taken from either a finger stick or a vein in the arm to check the sugar level. An injection of a small amount of a radioactive drug called FDG ( [F18] fluorodeoxyglucose) which is a chemical similar to sugar will be administered into a vein in the arm or hand. Approximately 45 to 60 minutes after the injection of FDG, the patient will be asked to urinate (to empty the bladder).

The patient will be set up in the PET/CT scanner using a vacuum cushion for immobilization in the supine position with feet tied and hands across the chest or above the head. There will also be a respiration-monitoring device called a marker block placed 5cm below the patient's xyphoid process. An infrared camera at the foot of the CT table will capture the images of the marker block and relay them to the RPM computer, which in turn will translate the images into a respiratory pattern. The audio coach (which instructs the patient in regulating breathing) will be calibrated to both patient comfort and time of expiration, inspiration, and full breathing cycle. The placing of the patient in a body immobilization device will take about 10-15 minutes. The patient will need to lie still for about 30 minutes before the completion of the 4D PET scan. The PET/CT scanner will then be programmed to acquire a retrospective 4D CT scan with a set of images for each phase of the breathing cycle. This scan will take place immediately after the PET scan. It will take around 5-10 minutes. The physician or physicist will then select the number of breathing phases to use while the software program selects the best image for each selected breathing phase.

The entire FDG-PET/CT scan procedure is expected to take about 2 hours.

Treatment Planning

Treatment planning will be carried out using the planning station for the radiosurgery equipment being used for treatment. The gross tumor volume (GTV) will be contoured on the fused image set. Two GTV volumes will be contoured; the gross tumor as seen on CT alone and the gross tumor corresponding to FDG avidity. No margins will be added for clinical target volume (CTV), but custom margins will be added for the planning target volume (PTV) based on the findings of the 4D FDG-PET/CT motion study assessment. The treatment will be prescribed to the isodose line that best covers the planning target volume, which will typically be the 80% isodose line.

Treatment Delivery

SBRT will take place within 14 days of the treatment planning scan. The planning data containing the coordinates of tumor isocenter, the external infrared markers, and the implanted markers are transferred to the appropriate platform depending on the treating machine. If the patient meets the criteria of gating technique then treatment delivery will be accomplished using the appropriate gating technology. Depending on the technology used external infrared markers attached to the patient's skin or a marker block placed on the patient's chest is used to determine the breathing pattern. The size of beam-on window will be determined based on the target motion as detected by the 4D FDG-PET/CT scan. The threshold for gated treatment delivery is determined based upon the target motion due to respiration.

The daily initial positioning during treatment delivery will be performed using lasers and skin marks and infrared optical markers as appropriate. The target isocenter will be verified using daily imaging. Depending on the platform used, the moving target will be positioned within the beam under infrared and/or image guidance

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* A life expectancy of at least 6 months with a Karnofsky performance status of at least 70
* The target lesion(s) can be accurately measured in at least one dimension according to RECIST and must have a maximum tumor volume of ≤ 100 cm3
* No prior radiotherapy to the upper abdomen
* Previous systemic chemotherapy or non-radiation local therapy (such as surgery, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) is allowed. The lesion must however have shown criteria of progression based on RECIST. Local therapy must be completed at least 4 weeks prior to the baseline scan. This is to create a safer treatment environment and to help determine the effect of treatment by SBRT alone. Patients will be allowed to go onto appropriate systemic therapy, as determined by their medical oncologist, 2 weeks following delivery of SBRT
* Patients with resectable disease will be eligible for participation if they have comorbidities precluding surgery or refuse to undergo an operation
* Cirrhotic status of Child-Pugh class A or B
* Patients can have extra-hepatic disease, provided the hepatic disease is the highest burden, the extra-hepatic disease is low burden and potentially treatable with surgery, ablative radiation therapy, or US Food and Drug Administration-approved first- or second-line systemic therapy regimens
* Patient's will have no evidence of gross vascular invasion.
* Patients will have no more than 3 distinct lesions, all being ≤ 3cm in greatest dimension, OR 1 lesion ≤ 6cm in greatest dimension
* Platelet count ≥ 60 x 109/L, Hemoglobin ≥ 8.5 g/dL, WBC ≥ 2000/μL International normalized ratio (INR) must be ≤ 2.3. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists
* Other baseline labs must meet the following criteria: total bilirubin < 3mg/dl, albumin> 2.5mg/dl, and liver enzymes less than three times the upper limit of normal. Creatinine must also be < 1.8mg/dl or a creatinine clearance > 50ml/min
* Must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts

Exclusion Criteria:

* Renal failure requiring hemo- or peritoneal dialysis
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 4.0), congestive heart failure (> New York Heart Association (NYHA) class 2), active coronary artery disease (CAD), cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin), uncontrolled hypertension and any condition which could jeopardize the safety of the patient and his/her compliance in the study . Myocardial infarction more than 6 months prior to study entry is permitted
* A history of variceal bleeding where the varices have not been eradicated or decompressed by shunt placement
* History of an active connective tissue disorder
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Pregnant or breast-feeding patients are excluded from this study because abdominal radiation therapy has potential for teratogenic and/or abortifacient effects
* Portal vein occlusion
* Extensive liver tumor burden, defined as more than 75% of the liver.
* Patients with primary tumor histology of lymphoma, leukemia, or germ cell tumor
* Patients with hepatocellular carcinoma will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03-23 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Ellsworth, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center - Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT - 50 Gy: Stereotactic Body Radiation Therapy: SBRT:
  Patients received 50 Gy in 5 fractions (10 Gy/fx) delivered over a 2-week period.
- SBRT - 60 Gy: Stereotactic Body Radiation Therapy: SBRT:
  Patients received 60 Gy in 5 fractions (12 Gy/fx) delivered over a 2-week period.
Period: 50 Gy
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: 60 Gy
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Started | 0 | 6
Completed | 0 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Median (Full Range); unit: years] | 66.0 [56.0 to 75.0] | 68.0 [53.0 to 81.0] | 66.0 [53.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Score [Number; unit: participants] — 0 = Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1 = Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature). 2 = Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities) 3 = Symptomatic, >50% in bed, but not bedbound (Limited self-care) 4 = Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair) 5 = Death
  participants
    ECOG = 1 | 1 | 0 | 1
    Unknown | 2 | 6 | 8
Karnofsky Score of Performance Status [Number; unit: participants] — 100% Normal; no complaints or evidence of disease. 90% Can do normal activity; minor signs of disease.80% Normal activity with effort; some signs of disease.70% Cares for self. Unable to do normal activity / active work.60% Needs occasional assistance, but able to care for most needs.50% Requires considerable assistance/frequent medical care. 40% Disabled; requires special care/assistance.30% Severely disabled; hospitalization indicated although death not imminent. 20% Very sick; hospitalization needed; active supportive necessary. 10% Moribund; fatal processes progressing rapidly. 0% Dead.
  participants
    Karnofsky Score = 70 | 1 | 1 | 2
    Karnofsky Score = 90 | 0 | 5 | 5
    Karnofsky Score = 100 | 1 | 0 | 1
    Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD as determined by dose limiting toxicities (DLT), defined as any grade III stomach, bowel, liver, or spinal cord toxicity, or any grade IV toxicity per RTOG criteria. Only toxicities observed prior to 7 months after the last fraction of radiation were considered. The MTD is the highest dose level at which no more than 1 of 6 treated patients experiences a DLT.
Time Frame: Up to 16 Months
Population: All patients that received study treatment.
Measure: Number; unit: Gy
Groups:
- All Participants: Stereotactic Body Radiation Therapy (SBRT) Patients that received at least one dose of either 50 Gy or 60 Gy in 5 fractions (12 Gy/fx) delivered over a 2-week period.
Arm/Group | All Participants
Number analyzed (Participants) | 9
Gy | 60

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: Dose limiting toxicity (DLT) will be defined as any grade III stomach, bowel, liver, or spinal cord toxicity, or any grade IV toxicity as defined by the Radiation Therapy Oncology Group (RTOG).
Time Frame: Up to 16 Months
Population: All patients that received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

3. Secondary Outcome: Local Control
Description: Proportion of treated patients with stable disease (SD), partial response (PR), or complete response (CR) in the target lesion(s) per Response Evaluation Criteria in Solid Tumors (RECIST) in the target lesion(s) at one-year post-treatment. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. All lymph nodes must be non-pathological in size (<10mm short axis); PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 6 years and 4 months (study population)
Population: All patients treated per protocol and radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 2 | 6
Participants
  Complete Response | 1 | 1
  Partial Response | 0 | 3
  Stable Disease | 1 | 1

4. Secondary Outcome: Local Response Rate
Description: Proportion of patients who experience local partial response (PR), or complete response (CR) in the target lesion(s) per Response Evaluation Criteria in Solid Tumors (RECIST) at any point in the first year of follow-up. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis); PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 6 years and 4 months (study population)
Population: All patients treated per protocol and radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 2 | 6
Participants
  Complete Response | 1 | 1
  Partial Response | 0 | 3

5. Secondary Outcome: FACT-G - Health Related Quality of Life (HRQL) Over Time
Description: Health related quality of life associated with this SBRT will be assessed over time using the FACT-G assessment tool, a self-administered questionnaire that measures quality of life within the prior 7 days in patients being treated for cancer. The tool has 27 items with a 5-point Likert-type scale, (0 = Not at all to 5 = Very Much). Subscales include Physical Well-Being max score=28), Social/Family Well-Being (max score=28), Emotional Well-Being (max score=24), Functional Well-Being (max score=28). Total scores range from 0 to 108. Questions are phrased so that higher numbers indicate a better health state, with some items reverse-scored.
Time Frame: 1-2 months, 3-5 months, 6-8 months, 9-11 months,12-14 months,15-17 months, 18-20 months, 21-23 months, 24-26 months
Population: All treated patients that completed QoL surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 3 | 6
score on a scale
  Screening: number analyzed (Participants) | 3 | 4
  Screening | 90.3 (15.0) | 88.0 (16.3)
  Initial Rx Therapy: number analyzed (Participants) | 2 | 4
  Initial Rx Therapy | 82.6 (35.9) | 82.5 (23.0)
  Post completion of RX Therapy: number analyzed (Participants) | 1 | 3
  Post completion of RX Therapy | 107.0 | 91.0 (14.7)
  1-2 months post final Rx: number analyzed (Participants) | 2 | 5
  1-2 months post final Rx | 69.0 (5.7) | 78.0 (20.9)
  3-5 months post final Rx: number analyzed (Participants) | 2 | 6
  3-5 months post final Rx | 86.5 (6.4) | 83.1 (17.4)
  6-8 months post final Rx: number analyzed (Participants) | 1 | 4
  6-8 months post final Rx | 87.0 | 85.1 (17.0)
  9-11 months post final Rx: number analyzed (Participants) | 0 | 4
  9-11 months post final Rx |  | 80.4 (21.7)
  12-14 months post final Rx: number analyzed (Participants) | 0 | 4
  12-14 months post final Rx |  | 84.7 (16.1)
  15-17 months post final Rx: number analyzed (Participants) | 0 | 1
  15-17 months post final Rx |  | 71.0
  18-20 months post final Rx: number analyzed (Participants) | 2 | 2
  18-20 months post final Rx | 78.0 (0.0) | 74.5 (17.7)
  21-23 months post final Rx: number analyzed (Participants) | 0 | 2
  21-23 months post final Rx |  | 69.0 (9.9)
  24-26 months post final Rx: number analyzed (Participants) | 0 | 1
  24-26 months post final Rx |  | 69.0

6. Secondary Outcome: Functional Assessment of Cancer Therapy-Hepatobiliary Index (FSHI) Over Time
Description: Functional Assessment of Cancer Therapy-Hepatobiliary Index (FSHI) subscale was used to assess health-related quality of life associated with SBRT. The FACT-Hep is part of the Functional Assessment of Chronic Illness Therapy (FACIT; 13) measurement system and includes the FACT-General (FACT-G) and an 8-item module specifically designed for patients diagnosed with hepatobiliary carcinomas.
  FACT-Hep questions are scored using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much), with overall scores ranging from 0-32.
  Questions are phrased so that higher numbers indicate a better health state, with some items reverse-scored.
Time Frame: 1-2 months, 3-5 months, 6-8 months, 9-11 months,12-14 months,15-17 months, 18-20 months, 21-23 months, 24-26 months
Population: All patients on study that completed QoL surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 3 | 6
score on a scale
  Screening: number analyzed (Participants) | 3 | 4
  Screening | 27.0 (5.0) | 27.2 (4.6)
  Initial Rx Therapy: number analyzed (Participants) | 2 | 4
  Initial Rx Therapy | 29.5 (3.5) | 24.5 (8.2)
  Post completion of RX Therapy: number analyzed (Participants) | 1 | 3
  Post completion of RX Therapy | 31.0 | 25.3 (5.8)
  1-2 months post final Rx: number analyzed (Participants) | 2 | 5
  1-2 months post final Rx | 24.5 (2.1) | 21.2 (7.7)
  3-5 months post final Rx: number analyzed (Participants) | 2 | 6
  3-5 months post final Rx | 25.0 (0.0) | 24.3 (5.8)
  6-8 months post final Rx: number analyzed (Participants) | 1 | 3
  6-8 months post final Rx | 29.0 | 26.7 (4.6)
  9-11 months post final Rx: number analyzed (Participants) | 0 | 4
  9-11 months post final Rx |  | 24.2 (5.7)
  12-14 months post final Rx: number analyzed (Participants) | 0 | 4
  12-14 months post final Rx |  | 24.2 (4.6)
  15-17 months post final Rx: number analyzed (Participants) | 0 | 1
  15-17 months post final Rx |  | 18.0
  18-20 months post final Rx: number analyzed (Participants) | 1 | 2
  18-20 months post final Rx | 23.0 | 22.0 (4.2)
  21-23 months post final Rx: number analyzed (Participants) | 0 | 2
  21-23 months post final Rx |  | 22.5 (0.7)
  24-26 months post final Rx: number analyzed (Participants) | 0 | 1
  24-26 months post final Rx |  | 21.0

7. Secondary Outcome: FACT-Hep-Trial Outcome Index (TOI)
Description: Trial Outcome Index (TOI), the sum of the physical and functional well-being subscales and the additional concerns subscale is calculated. The TOI is a commonly used endpoint in clinical trials because it is responsive to change, whereas the social/family and emotional well-being subscale scores do not change as quickly over time or have as great of change subsequent to pharmacological treatment. The FACT-Hep is part of the Functional Assessment of Chronic Illness Therapy (FACIT 13) measurement system and includes the FACT-General (FACT-G) and an 18-item module specifically designed for patients diagnosed with hepatobiliary carcinomas with domain scores ranging from 0-32. FACT-Hep questions are scored using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Total Index scores range from 0 to 128. Higher scores are associated with better QoL or fewer symptoms.
Time Frame: 1-2 months, 3-5 months, 6-8 months, 9-11 months,12-14 months,15-17 months, 18-20 months, 21-23 months, 24-26 months
Population: All patients on study that completed QoL surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
Number analyzed (Participants) | 3 | 6
score on a scale
  Screening: number analyzed (Participants) | 3 | 4
  Screening | 108.3 (13.7) | 106.0 (17.6)
  Initial Rx therapy session: number analyzed (Participants) | 2 | 4
  Initial Rx therapy session | 107.0 (25.5) | 98.5 (29.0)
  After completion of final Rx: number analyzed (Participants) | 1 | 3
  After completion of final Rx | 126.0 | 104.0 (21.4)
  01-02 months post final Rx: number analyzed (Participants) | 2 | 5
  01-02 months post final Rx | 92.5 (10.6) | 90.4 (27.2)
  03-05 months post final Rx: number analyzed (Participants) | 2 | 6
  03-05 months post final Rx | 101.0 (4.2) | 92.5 (16.3)
  06-08 months post final Rx: number analyzed (Participants) | 1 | 3
  06-08 months post final Rx | 117.0 | 106.0 (14.8)
  09-11 months post final Rx: number analyzed (Participants) | 0 | 4
  09-11 months post final Rx |  | 94.0 (24.8)
  12-14 months post final Rx: number analyzed (Participants) | 0 | 4
  12-14 months post final Rx |  | 99.8 (20.1)
  15-17 months post final Rx: number analyzed (Participants) | 0 | 1
  15-17 months post final Rx |  | 73.5
  18-20 months post final Rx: number analyzed (Participants) | 1 | 2
  18-20 months post final Rx | 103.0 | 85.0 (18.4)
  21-23 months post final Rx: number analyzed (Participants) | 0 | 2
  21-23 months post final Rx |  | 83.5 (6.4)
  24-26 months post final Rx: number analyzed (Participants) | 0 | 1
  24-26 months post final Rx |  | 83.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of up to 5 years.
Arm/Group | SBRT - 50 Gy | SBRT - 60 Gy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 2/3 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT - 50 Gy (N=3) | SBRT - 60 Gy (N=6)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 4
Hepatobiliary disorders - Other, specifyLDH increased (Hepatobiliary disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Investigations - Other, specifyedema in lower extremities (Investigations) | 1 | 0
Investigations - Other, specifyLDH increased (Investigations) | 0 | 1
Investigations - Other, specifyRib pain (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyErythema-right breast (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT01360606/Prot_SAP_000.pdf